CLINICAL TRIAL: NCT03983434
Title: Fecal Bile Acids, Fecal Short Chain Fatty Acids and the Intestinal Microbiota in Patients With Irritable Bowel Syndrome (IBS) and Control Volunteers: Diet Challenge
Brief Title: Irritable Bowel Syndrome and Control Volunteers: Diet Challenge
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study physician left the university
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Huiping Xu, Associate Professor, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1903209172; K23DK122015 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: microbiome; microbiota; short chain fatty acids; prebiotic; bile acids
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): Adults ages 18-65 years with no prior history of gastrointestinal diseases or symptoms.
  Interventions: Dietary Supplement: Inulin
- Irritable Bowel Syndrome Patients with Diarrhea (Experimental): Patients with irritable bowel syndrome (IBS) with diarrhea, ages 18-65 years fulfilling Rome IV criteria for IBS
  Interventions: Dietary Supplement: Inulin
- Irritable Bowel Syndrome Patients with Constipation (Experimental): Patients with irritable bowel syndrome (IBS) with constipation, ages 18-65 years fulfilling Rome IV criteria for IBS
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin ingestion is not being used to diagnose, treat, or prevent IBS. Inulin is being used to study an individual's ability to ferment dietary fiber.

SUMMARY:
The purpose of this study is to study the relationship between the bile acids, short chain fatty acids and bacteria within the intestines. The hypothesis is that changes in the bacterial composition of the stool are associated with the differences in bile acids and short chain fatty acids in patients having irritable bowel syndrome compared to healthy individuals.

DETAILED DESCRIPTION:
The Study involves 3 visits and will in include 3 types of subjects - those who have irritable bowel syndrome (IBS) with constipation (IBS-C), IBS with diarrhea (IBS-D) and those who have no IBS symptoms or diagnosis.

Visit 1

* Volunteers will read and sign this informed consent after all questions about the study have been answered
* This is a screening visit and we may determine that volunteers ineligible to continue to participate in the study.
* Volunteers will have a medical history taken including demographics, history of symptoms and illness
* Volunteers will be asked about all medications
* A physical exam will be performed by the physician.
* Vital signs will be measured.
* Urine Pregnancy test may be done for woman in the reproductive age range.
* Eligible participants will be provided with a take-home lasagna meal.
* Participants will be given instructions and supplies for collection, storage and transportation of stool for the next visit.
* Participants will be provided with instructions for a low fiber, high fat diet which should be consumed for 2 days before stool collection and during the 2 days of stool collection. Instructions will also come with materials to allow participants to record diet intake during these 4 days.
* Participants will be provided a bowel pattern diary to record bowel symptoms over the course of the study

Day 1: this may be the same as Visit 1 or it may be a different day. It will depend upon the day that participants can make it back to the clinic for the Day 5 visit.

Day 2-4 (at home):

* Participants record stool symptoms and patterns in a diary daily starting from Day 2 to Day 5.
* During this time, participants will be instructed to consume a low fiber diet, avoid alcohol, and start a 4-day 100 g fat diet.
* On the evening before Day 5, a standardized, completely digestible, and non-fermentable meal (lasagna) will be consumed which will be provided to you on Day 1.
* Participants will collect stool at home on Day 4 and 5 and store as per instructions provided on Visit 1. They will

Day 5 (Visit 2):

* Participants return to the clinic on Day 5 after an overnight fast.
* You will receive a standard breakfast and lasanga meal with 10 g inulin (Orafti®) powder and 200 mL of water.
* Take-home meals will be provided (white bread sandwich with ham or cheese) to be consumed at 4 and 8 hours after breakfast.

Day 6 (Visit 3):

* Participants will return to the clinic in order to return stool collections and the daily diaries.
* Participants may also submit diaries by fax or email.

Day 30-90

• Optional dietary follow-up (Day 30-90): To further assess the utility of the 24 hour dietary recall, willing participants will be invited to participate in a an optional follow-up activity during which they will complete the Automated Self-Administered Dietary Assessment Tool with or without assistance of a trained interviewer. Interested volunteers will be contacted by phone and provided instructions on how to complete the tool online by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS, ages 18-65 fulfilling Rome IV criteria and asymptomatic controls with no prior history of GI disease or symptoms.
* Participants should be on a stable and consistent diet regimen and should not be following an extreme diet intervention such as gluten-free or a low FODMAP diet at the time of study participation.

Exclusion Criteria:

* Participants with microscopic/lymphocytic/collagenous colitis, inflammatory bowel disease, celiac disease, visceral cancer, chronic infectious disease, immunodeficiency, uncontrolled thyroid disease, history of liver disease or history of elevated AST/ALT > 2.0x the upper limit of normal
* Prior radiation therapy of the abdomen or abdominal surgeries except for C-section, tubal ligation, vaginal hysterectomy and appendectomy or cholecystectomy, > 6 months prior to study initiation.
* Ingestion of any prescription, over the counter, or herbal medications which can affect GI transit or study interpretation (e.g. opioids, narcotics, anticholinergics, norepinephrine reuptake inhibitors, nonsteroidal anti-inflammatory drugs, COX-2 inhibitors, bile acid sequestrants) within 6 months of study initiation for asymptomatic volunteers or within 2 days before study initiation for IBS patients. Rescue therapy to facilitate stool collection will be permitted where needed.
* Any females who are pregnant or trying to become pregnant or breast-feeding
* Antibiotic usage within 3 months prior to study participation
* Prebiotic or probiotic usage within the 2 weeks prior to study initiation
* Regular use of tobacco products within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huiping XU, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Started | 17 | 3 | 9
Completed | 16 | 2 | 6
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea | Total
Number analyzed (Participants) | 17 | 3 | 9 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 3 | 9 | 28
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (14.9) | 26.4 (6) | 36.1 (9.5) | 35.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 7 | 21
  Male | 5 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 3 | 9 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 0 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 8 | 2 | 8 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Fecal Bile Acids
Description: Stool samples will be collected over 2 days for measurement of fecal bile acids (mcmol/48h) by high performance liquid chromatography-mass spectometry
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: mcmol/48 hours
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 2 | 6
mcmol/48 hours | 471.5 [331.5 to 612.5] | 347 [159 to 535] | 329.5 [145 to 515]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = .62, Kruskal-Wallis

2. Primary Outcome: Total Fecal Short Chain Fatty Acids
Description: Stool samples will be collected for measurement of measurement of short chain fatty acids (mmol/kg) by liquid chromatography-mass spectrometry
Time Frame: 48 hours
Population: One subject in the group of Irritable Bowel Syndrome Patients with Constipation had missing data in short chain fatty acids.
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 1 | 6
mmol/kg | 359.8 [233.1 to 473.2] | 157.1 [157.1 to 157.1] | 276.9 [168.6 to 408.1]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.17, Kruskal-Wallis

3. Primary Outcome: Individual Fecal Short Chain Fatty Acids - Acetate
Description: as for outcome 2
Time Frame: 48 hours
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 1 | 6
mmol/kg | 255.7 [147.5 to 300.1] | 113.9 [113.9 to 113.9] | 202.5 [121.7 to 266]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.17, Kruskal-Wallis

4. Primary Outcome: Individual Fecal Short Chain Fatty Acids - Propionate
Description: as for outcome 2
Time Frame: 48 hours
Population: One subject in the group of Irritable Bowel Syndrome Patients with Constipation had missing short chain fatty acids
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 6 | 1
mmol/kg | 59.7 [39.8 to 86] | 22.8 [22.8 to 22.8] | 39.1 [25.3 to 51.1]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.079, Kruskal-Wallis

5. Primary Outcome: Individual Fecal Short Chain Fatty Acids - Butyrate
Description: as for outcome 2
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: mmol/kg
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 1 | 6
mmol/kg | 57.5 [29.1 to 70.2] | 20.5 [20.5 to 20.5] | 37.6 [16.9 to 91]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.47, Kruskal-Wallis

6. Primary Outcome: Fecal Microbial Population
Description: Stool samples will be be collected from participants for nucleic acid extraction, shotgun sequencing is used to measure microbial communities and profiles of specimens. Shannon index is calculated to measure the diversity of species. The minimum value is 0. There is no upper limit. The higher the Shannon index is, the greater the diversity of species is.
Time Frame: 48 hours
Population: Microbiome sequencing was completed on all collected specimens.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 0 | 7
units on a scale | 3 [2.75 to 3.5] |  | 3.6 [3.2 to 3.8]

7. Primary Outcome: Fecal Inulin
Description: Fecal inulin content will be measured using short acid hydrolysis and high-performance liquid chromatography
Time Frame: 48 hours
Population: Measures of inulin evolved over time and many subjects did not have inulin measured as a fraction.
Measure: Median (Inter-Quartile Range); unit: % of fructose from inulin/total fructose
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 7 | 0 | 3
% of fructose from inulin/total fructose | 3.6 [0.8 to 5.4] |  | 17.1 [7.4 to 25]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.03, Kruskal-Wallis

8. Secondary Outcome: Percent Primary Fecal Bile Acids
Description: Stool samples will be collected over 2 days for measurement of fecal bile acids (mcmol/48h) by high performance liquid chromatography-mass spectrometry. Percent primary bile acids is then calculated as primary bile acids divided by total bile acids multiplied by 100.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: % of primary/total fecal bile acids
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 2 | 6
% of primary/total fecal bile acids | 2.7 [1 to 26.8] | 0.4 [0.3 to 0.5] | 2.1 [0.6 to 10.3]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.14, Kruskal-Wallis

9. Secondary Outcome: Stool Characteristics - Stool Frequency in 4 Days
Description: Stool characteristics will be measured using a 4 day bowel diary. Stool frequency is the total number of bowel movements in 4 days summarized on the subject level.
Time Frame: 4 days
Measure: Median (Inter-Quartile Range); unit: Number of bowel movements in 4 days
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 2 | 6
Number of bowel movements in 4 days | 4.5 [4 to 5.5] | 0.5 [0 to 1] | 5 [2 to 10]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.074, Kruskal-Wallis

10. Secondary Outcome: Stool Characteristics - Stool Form
Description: Stool characteristics will be measured using a 4 day bowel diary. Stool form is on a scale from 1 to 7, where 1=hard lumps, 2=lumps sausage,3=cracked sausage, 4=normal, 5=soft lumps, 6=mushy,7=watery, summarized on the level of bowel movements.
Time Frame: 4 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Bowel movements
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 2 | 6
Number analyzed (Bowel movements) | 73 | 1 | 33
score on a scale | 4 [3 to 5] | 1 [1 to 1] | 5 [4 to 6]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other; p = 0.004, Kruskal-Wallis

11. Secondary Outcome: Stool Characteristics - Ease of Passage
Description: Stool characteristics will be measured using a 4 day bowel diary. Ease of passage is on a scale from 1 to 7, where 1=manual disimpaction, 2=enema needed, 3=straining needed, 4=normal, 5=urgent without pain, 6=urgent with pain, 7=incontinent, also summarized on the level of bowel movements.
Time Frame: 4 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Bowel movements
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 16 | 2 | 6
Number analyzed (Bowel movements) | 73 | 1 | 33
score on a scale | 4 [4 to 4] | 3 [3 to 3] | 4 [4 to 5]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other; p = 0.17, Kruskal-Wallis

12. Other Pre Specified Outcome: Energy
Description: Optional 24-hour dietary intake will be submitted using web-based Automated Self-Administered Dietary Assessment Tool developed by the National Cancer Institute (https://epi.grants.cancer.gov/asa24/). Dietary intake within a 24-hour period in 30-90 days after study enrollment were collected.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
Number analyzed (Participants) | 12 | 2 | 6
kcal | 1887.6 [1563.9 to 2507.5] | 2083.8 [1801.3 to 2366.4] | 2246.4 [1540.1 to 2509.8]
Statistical Analysis 1: Comparison: Healthy Volunteers vs Irritable Bowel Syndrome Patients With Constipation vs Irritable Bowel Syndrome Patients With Diarrhea; Test type: Other — Due to the skewness of the data, outcome measures were summarized using median and interquartile range; p = 0.98, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Healthy Volunteers | Irritable Bowel Syndrome Patients With Constipation | Irritable Bowel Syndrome Patients With Diarrhea
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/16 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03983434/Prot_SAP_000.pdf